CLINICAL TRIAL: NCT05703438
Title: The Effect of a Nutritionally Balanced Low Calorie Diet Based on Traditional Indonesian Foods on Obese People's Metabolic Biomarkers
Brief Title: The Effect of a Low-calorie Diet With Balanced Nutrition on Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andalas University (Other)
Collaborators: Universitas Sumatera Utara (Other); Hasanuddin University (Other)
Responsible Party: Principal Investigator, Nur Indrawaty Lipoeto, Clinical Professor, Andalas University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RKI2022
Record Dates: First submitted 2022-12-05; First posted 2023-01-30 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Metabolic Syndrome, Protection Against
Keywords: Nutritionally balanced low-calorie diet; Archipelago diet; Metabolic biomarkers
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The study was conducted by providing a daily calorie deficit of 500-600 kcal to the usual intake of each participant. The study was conducted for 8 weeks. Examination of metabolic biomarkers is carried out before and after the diet intervention is administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritionally balanced low-calorie diet (Experimental): Experimental study with pre and post design
  Interventions: Other: Nutritionally balanced low-calorie diet

INTERVENTIONS:
Other: Nutritionally balanced low-calorie diet — Dietary interventions were given with a calorie deficit of 500-600 kcal from the participants' usual daily intake.

SUMMARY:
The study looked at how a nutritionally balanced low-calorie diet based on traditional Indonesian foods affected obese people's metabolic biomarkers. The traditional Indonesian foods presented here are Minangkabau cuisine. Body mass index, waist circumference, systolic and diastolic blood pressure, body fat mass percentage, fasting blood sugar levels, and lipid profiles are among the metabolic biomarkers measured. The provision of a balanced nutritionally low-calorie diet based on traditional Indonesian foods, according to the researchers, will have a significant effect on the metabolic biomarkers of obese people.

DETAILED DESCRIPTION:
The research was carried out at RSUP dr. M. Djamil Padang. The research ethics commission of Andalas University's Faculty of Medicine granted the study an ethical permit. Health workers with a BMI of more than 25 kg/m2 became the study population, and officers who agreed to participate in the study after filling out the informed consent form were included in the study. There were 91 people in the study. The study lasted eight weeks (56 days). A week before the study, participants were interviewed about their daily intake using 24-hour food recall, and anthropometric measurements were taken using calibrated tools and performed by trained officers.

Subjects underwent a one-week pre-treatment period (baseline period, beginning on D-day 6 and ending on D-day 0), during which they were asked not to take any supplements. All participants had their anthropometric measurement, blood pressure, body fat percentage, fasting blood sugar levels, and lipid profile checked on day 0 and day 57.

The Nutrisurvey 2005 application was used to process the daily intake of participants obtained from a 24-hour food recall interview. Dietary interventions were given with a calorie deficit of 500-600 kcal from the participants' usual daily intake. A Minangkabau food menu is provided as part of the diet. Participants are given a list of daily menus, which include breakfast, lunch, and dinner. Researchers provided lunch for study participants, while breakfast and dinner were prepared independently by participants using the dietary guidelines and menus provided. Participants kept a food diary, which was collected and evaluated twice a week. The research team also controls and motivates all participants via Whatsapp groups. The study's findings were analyzed using the SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Employee of RSUP dr. M. Djamil, Padang who suffers from obesity (BMI ≥ 25 kg / m2)
* Willing to follow the research by signing an informed concent

Exclusion Criteria:

* Did not come and could not be found at the time of research data collection
* Unable to follow the dietary arrangements as set
* Taking anti-diabetic or anti-lipid drugs
* Use of contraceptives or hormonal drugs
* In the treatment of radiotherapy or chemotherapyi

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline body mass index at 8 weeks. | up to 8 weeks
  A person's weight in kilograms divided by the square of height in meters
Change from baseline waist circumference at 8 weeks. | up to 8 weeks
  The measurement taken around the abdomen at the level of the umbilicus (belly button).
Change from baseline systolic and diastolic blood pressure at 8 weeks. | up to 8 weeks
  Measured using a digital sphygmomanometer
Change from baseline fat mass percentage at 8 weeks. | up to 8 weeks
  Measured using bioimpedance analysis (BIA)
Change from baseline fasting blood sugar levels at 8 weeks. | up to 8 weeks
  Measured using clinical chemistry analyzer
Change from baseline lipid profile levels at 8 weeks. | up to 8 weeks
  The lipid profile examined included total cholesterol, triglycerides, HDL (high density lipoprotein) cholesterol, and LDL (low density lipoprotein) cholesterol. Measured using clinical chemistry analyzer (photometer).

CONTACTS AND LOCATIONS:
Overall Officials: Nurindrawaty Lipoeto, PhD, Principal Investigator — Universitas Andalas
Locations (1):
- Universitas Andalas, Padang, West Sumatra, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Starting 6 months after publication for 1 year
Access Criteria: other researcher can contact us trough e-mail.

REFERENCES:
- [Background] Han TS, Lean ME. A clinical perspective of obesity, metabolic syndrome and cardiovascular disease. JRSM Cardiovasc Dis. 2016 Feb 25;5:2048004016633371. doi: 10.1177/2048004016633371. eCollection 2016 Jan-Dec. PMID 26998259
- [Result] Witjaksono F, Jutamulia J, Annisa NG, Prasetya SI, Nurwidya F. Comparison of low calorie high protein and low calorie standard protein diet on waist circumference of adults with visceral obesity and weight cycling. BMC Res Notes. 2018 Sep 21;11(1):674. doi: 10.1186/s13104-018-3781-z. PMID 30241565